CLINICAL TRIAL: NCT05304468
Title: Phase III Randomized Non-inferiority Trial of Reduced-dose Versus Standard Dose Radiotherapy for Stage II-III Nasopharyngeal Carcinoma Which Have Favorable Response After Induction Chemotherapy
Brief Title: Reduced-dose Versus Standard Dose Radiotherapy for Nasopharyngeal Carcinomain
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-017
Record Dates: First submitted 2022-03-28; First posted 2022-03-31 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; radiotherapy; induction chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Induction Chemotherapy

STUDY DESIGN:
Intervention Model Description: phase III non-inferiority
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced-dose group (Experimental): After 2 cycles of induction chemotherapy, patients with favorable response undergo low-dose (60Gy) intensity-modulated radiotherapy (IMRT) 5 days per week for approximately 6 weeks (30 fractions). Patients also receive concurrent cisplatin once every three weeks for 2 cycles.
  Interventions: Radiation: IMRT; Drug: induction chemotherapy; Drug: cisplatin concurrent chemotherapy
- Standard dose group (Active Comparator): After 2 cycles of induction chemotherapy, patients with favorable response undergo standard-dose (70Gy) intensity modulated radiotherapy (IMRT) 5 days per week for approximately 7 weeks (33 fractions). Patients also receive concurrent cisplatin once every three weeks for 3 cycles.
  Interventions: Radiation: IMRT; Drug: induction chemotherapy; Drug: cisplatin concurrent chemotherapy

INTERVENTIONS:
Radiation: IMRT — Patients in experimental group received reduced dose IMRT
Drug: induction chemotherapy — cisplatin-based induction chemotherapy for two cycles
Drug: cisplatin concurrent chemotherapy — cisplatin 100mg/m2, for two(60Gy) or three cycles(70Gy)

SUMMARY:
To study the 2-year PFS (progression-free survival) of patients with stage II-III nasopharyngeal carcinoma treated with induction chemotherapy followed by two different doses of intensity modulated radiation therapy plus concurrent cisplatin chemotherapy

DETAILED DESCRIPTION:
To explore the 2 year PFS of patients with stageII-III nasopharyngeal carcinoma treated with induction chemotherapy followed by reduced-dose radiotherapy and cisplatin versus standard dose radiotherapy plus cisplatin concurrent chemotherapy. The enrolled patients will receive 2 cycles of cisplatin-based induction chemotherapy, if radiographic CR/PR and EBV DNA=0 after induction chemotherapy, the patients will be randomised assigned to received 60 Gy IMRT combined with 2 cycles of cisplatin concurrent chemotherapy or 70Gy IMRT combined with 3 cycles of cisplatin concurrent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients newly diagnosed with histologically confirmed non-keratinizing NPC (WHO type II or III).
2. Stage II-III（8thAJCC/UICC staging system)
3. Aged 18-70 years
4. ECOG = 0-1
5. HGB≥90 g/L，WBC≥4×109 /L，PLT≥100×109 /L
6. ALT,AST<1.5 x ULN；TBIL<1.5×ULN
7. CCR≥60ml/min or Cr<1.5×ULN
8. CR/PR and EBVDNA undetectable after induction chemotherapy
9. Signed informed consent

Exclusion Criteria:

1. WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma
2. Age <18 or >70years
3. Treatment with palliative intent
4. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer
5. Pregnancy or lactation
6. History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume)
7. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes
8. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2029-10-29 (Estimated)

PRIMARY OUTCOMES:
PFS (progression-free survival) | 2 year
  Defined as the time from randomization to documented disease recurrence (either distant metastasis or locoregional disease recurrence) or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival(OS) | 2 year
  Defined as the time from randomization to death from any cause
Locoregional relapse-free survival(LRFS) | 2 year
  Defined as the time from randomization to the first local or regional recurrence, or death from any cause.
  follow-up visit.
Distant metastasis-free survival(DMFS) | 2 year
  Defined as the time from randomization to the first distant metastasis or death from any cause.
Overall response rate | 3 months
  Tumour response rate was classified according to RECIST, version 1.1
Incidence rate of adverse events (AEs) | 2 year
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
Change of QoL | 1 year
  QoL scores were assessed for each scale by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) before induction chemotherapy, before radiotherapy, at the end of radiotherapy, at 3 months after radiotherapy, at 6 months after radiotherapy and 12 months after radiotherapy
Change of EORTC quality of life questionnaire(QLQ) Head and Neck score | 1 year
  QoL scores were assessed by using EORTC quality of life questionnaire(QLQ) Head and Neck. The QLQ-H&N35 is composed of seven multi-item symptom scales (pain, swallowing, sensation, speech, eating from a social,perspective, social interactions, and sexuality) and 11 single-item symptom scales (teeth, opening mouth,dry mouth, sticky saliva,coughing, felt ill, pain medication use, nutritional supplementation, feeding tube requirement, weight loss, and weight gain). All of the scales and items ranged in score from 0 to 100. A high score for a functional or global QoL scale represents a relatively high/healthy level of functional or global QoL, whereas a high score for a symptom scale or item represents a high number of symptoms or problems.All of the scores mentioned above were assessed at the below time point:before induction chemotherapy, before radiotherapy, at the end of radiotherapy, at 3 months after radiotherapy, at 6 months after radiotherapy and 12 months after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hai Qiang Mai, Dr, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen Universitty Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided